CLINICAL TRIAL: NCT02672215
Title: The Effectiveness of a Web-based Computer-tailored Intervention on Workplace Sitting: a Randomized Controlled Trial
Brief Title: RCT Computer-tailored Intervention on Workplace Sitting
Acronym: StartToStand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: EC/2012/320
Record Dates: First submitted 2016-01-20; First posted 2016-02-03 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- tailored group (Experimental): Received a web-based computer-tailored intervention including personalized feedback and tips on how to reduce and/or interrupt workplace sitting.
  Interventions: Behavioral: Start to stand
- generic group (Active Comparator): Received a web-based intervention containing generic information and tips to reduce and/or interrupt workplace sitting.
  Interventions: Behavioral: generic advice
- control group (No Intervention): A waitlist control condition and received the generic intervention after completing all measurements

INTERVENTIONS:
Behavioral: Start to stand — web-based computer-tailored intervention including personalized feedback and tips on how to reduce and/or interrupt workplace sitting
  Arms: tailored group
Behavioral: generic advice — general, non-tailored web-based generic advice with tips
  Arms: generic group

SUMMARY:
A theory-driven, web-based, computer-tailored advice to influence sitting at work was developed. The study investigated the effects of this computer-tailored intervention to influence workplace sitting on behavioural measures.

DETAILED DESCRIPTION:
The study investigated the effects of the theory-driven, web-based, computer-tailored intervention to influence workplace sitting on objectively measured sitting time, standing time and breaks from sitting, as well as self-reported context-specific sitting. The computer-tailored advice was compared to a generic advice and a 'no-advice' control at 1-month and 3-months follow-up. The 'tailored' group received a web-based computer-tailored intervention including personalized feedback and tips on how to reduce and/or interrupt workplace sitting. The 'generic' group received a web-based intervention containing generic information and tips to reduce and/or interrupt workplace sitting. The control group was a waitlist control condition and received the generic intervention after completing all measurements. Participants were recruited from a convenience sample of two companies (university and environmental agency) in Flanders (i.e. northern Dutch-speaking part of Belgium), mainly employing desk-based workers, having more than 100 staff members and each having at least three different worksite locations.

ELIGIBILITY:
Inclusion Criteria:

* being employed

Exclusion Criteria:

* not being able to stand

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1061 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
sitting time | one week
  objectively measured sitting time with ActivPAL
self-reported context-specific sitting time | one week
  self-reported context-specific sitting time with WSQ questionnaire
standing time | one week
  objectively measured standing time with ActivPAL
breaks from sitting | one week
  objectively measured breaks from sitting with ActivPAL

SECONDARY OUTCOMES:
psychosocial correlates of sitting | one week
  psychosocial correlates of sitting with questionnaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Cocker K, De Bourdeaudhuij I, Cardon G, Vandelanotte C. What are the working mechanisms of a web-based workplace sitting intervention targeting psychosocial factors and action planning? BMC Public Health. 2017 May 3;17(1):382. doi: 10.1186/s12889-017-4325-5. PMID 28468687
- [Derived] De Cocker K, De Bourdeaudhuij I, Cardon G, Vandelanotte C. The Effectiveness of a Web-Based Computer-Tailored Intervention on Workplace Sitting: A Randomized Controlled Trial. J Med Internet Res. 2016 May 31;18(5):e96. doi: 10.2196/jmir.5266. PMID 27245789